CLINICAL TRIAL: NCT06599528
Title: A Phase I Clinical Trial to Compare the Pharmacokinetics, Safety and Immunogenicity of SJ04 and Ovidrel® in Healthy Female Subjects in China
Brief Title: A Comparing Study Between SJ04 and Ovidrel® in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Centergene Pharmaceuticals Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SZSJ-SJ04-001
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Assisted Reproductive Technology; Female Infertility
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- T-R Group (Test-Reference drug) (Experimental): SJ04 is injected first and Ovidrel® is injected after 2-week period
  Interventions: Drug: T-R (Test-Reference drug)
- R-T Group(Reference-Test drug) (Experimental): Ovidrel® is injected first and SJ04 is injected after 2-week period
  Interventions: Drug: R-T (Reference-Test drug)

INTERVENTIONS:
Drug: T-R (Test-Reference drug) — T: SJ04 (Test drug) R: Ovidrel® (Referecne drug) 250 μg of SJ04 injection or Oviderl®, administered subcutaneously once at two week intervals.
  Arms: T-R Group (Test-Reference drug)
Drug: R-T (Reference-Test drug) — R: Ovidrel®(Referecne drug) T: SJ04 (Test drug) 250 μg of SJ04 or Oviderl®, administered subcutaneously once at two week intervals.
  Arms: R-T Group(Reference-Test drug)

SUMMARY:
This is a single-centre, randomised, open-label, single-dose, two-cycle, double-crossover study to compare the pharmacokinetics of SJ04 and Ovidrel® in healthy female subjects. Received a single subcutaneous injection administration of SJ04 Injection or Ovidrel®, both administered at a dose of 250 μg, once per cycle, and cross-administered after a washout period.

DETAILED DESCRIPTION:
SJ04 is a biosimilar of Ovidrel® and is highly similar to Ovidrel®. The purpose of this study was to evaluate the similarity of pharmacokinetics (PK) between recombinant human chorionic gonadotropin injection (SJ04) and Ovidrel® after administration by a single subcutaneous injection in healthy Chinese female subjects.

Forty-eight screened healthy female subjects were randomly divided into 2 groups, the T-R group and the R-T group, with 24 subjects in each group. On the morning of the day of administration, they received SJ04 injection or Ovidrel® single subcutaneous injection according to the randomisation table, both at a dose of 250 μg, once per cycle, and crossed over after a washout period.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female subjects aged 20 to 40 years old (including boundary values).
2. Weight not less than 45.0 kg, body mass index within the range of 19.0~26.0 kg/m2 (including boundary values).
3. Menstrual cycle regularity, or menstrual regularity before taking oral contraceptives (25-34 days, including boundary values).
4. The levels of follicle stimulating hormone(FSH), luteinizing hormone(LH), prolactin (PRL), estradiol (E2), progesterone (P), and testosterone (T) detected within 2-3 days after the last menstrual period before the first administration are within normal ranges or considered abnormal by the researchers to have no clinical significance.
5. LH levels <5 IU/L, FSH levels <4 IU/L at Day -1.

Exclusion Criteria:

1. Allergy or suspected allergy to any component of the experimental drug, control drug, GnRH, GnRH analogs used in this study.
2. Use of any LH preparation, human menopausal gonadotropin (hMG) or human chorionic gonadotropin (hCG) preparation within 3 months prior to screening.
3. Previously or currently suffering from the following diseases: hypothalamic or pituitary tumors, unexplained ovarian enlargement or cyst, Abnormal uterine bleeding of unknown etiology, malignant tumors of the ovaries, uterus, or breast, active thromboembolic diseases, uncontrollable thyroid or adrenal dysfunction, endocrine disorders such as hyperprolactinemia, polycystic ovary syndrome, ovarian hyperstimulation syndrome (OHSS), and ovarian dysfunction, other malignant tumors or diseases of the hypothalamus, pituitary gland, ovaries, and uterus (excluding uterine fibroids).
4. Ectopic pregnancy within 3 months prior to screening.
5. Presence of clinically significant acute or chronic infection at screening or enrolment。
6. Presence of localised disease affecting the hypodermic site, or inability to tolerate hypodermic injections。
7. Difficulty in blood collection or inability to tolerate venipuncture, or history of needle or blood sickness.
8. Prescription medications taken within 14 days or 5 half-lives prior to screening or over-the-counter medications (including proprietary and herbal medications) taken within 7 days or 5 half-lives prior to screening .
9. A history of chronic or serious illness or disease of the liver, kidneys, gastrointestinal tract, endocrine system, cardiovascular, neurological, metabolic, haematological, respiratory, or autoimmune systems or an existing disease of one of the above systems which, in the judgement of the investigator, makes him or her unsuitable for enrolment.
10. Abnormalities in vital signs, physical examination, laboratory tests (routine blood, blood biochemistry, urinalysis, coagulation, thyroid function), 12-lead electrocardiogram, liquid-based thin-layer cytometry (TCT), and ultrasound are judged by the investigator to be clinically significant and to warrant participation in the trial.
11. Positive tests for hepatitis B surface antigen, hepatitis C virus antibody, human immunodeficiency virus antibody, and syphilis spirochete antibody.
12. History of mental illness, substance abuse, drug dependence, or positive substance abuse screen (morphine, THC, methamphetamine, MDMA, ketamine) on the day of admission.
13. Excessive consumption of tea, coffee or caffeinated beverages in the 3 months prior to screening.
14. Drinking an average of more than 14 standard units of alcohol per week in the three months prior to screening, or inability to abstain from alcohol during the test period, or a positive breathalyser test result on the day of admission.
15. Smoke at least 5 cigarettes per day in the 3 months prior to screening or not be able to stop using any tobacco-based products during the trial.
16. Participated in a clinical trial of another drug within 28 days prior to screening and used the test drug, or participated in a clinical trial of a medical device within 1 month prior to screening.
17. History of blood donation or bleeding >400 ml within 3 months prior to screening.
18. During pregnancy or breastfeeding, or a positive pregnancy test result. The subject (or his/her partner) is planning to have children (including sperm and egg donation) throughout the trial period and for 3 months after the end of the trial. Unwilling to use one or more non-pharmacological contraceptive methods (e.g. total abstinence, condoms, ligation, etc.) during the trial period.
19. Subjects who withdrew from the trial for their own reasons and who, in the opinion of the investigator, were otherwise unsuitable to participate in the trial.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics: Area under the plasma concentration versus time curve (AUC) | day 8
  Analysis of equivalence of area under concentration-time curve from time 0 (predose) to the last quantifiable data point and to infinity of SJ04 and Ovidrel®
Pharmacokinetics: Peak Plasma Concentration (Cmax) | day 8
  Analysis of equivalence of Cmax of SJ04 and Ovidrel®

SECONDARY OUTCOMES:
Adverse events | day 8
  The Investigator will carefully monitor each subject throughout the study for any adverse events (coded to preferred term and system organ class using the Medical Dictionary for Regulatory Activities [MedDRA])
Immunogenicity | day 8
  antidrug antibodies (ADA) level

CONTACTS AND LOCATIONS:
Locations (1):
- Suzhou Municipal Hospital, Suzhou, Jiangsu, China